CLINICAL TRIAL: NCT04458987
Title: Identification and Validation of Addictology Expert Patients' Fields of Intervention With Inpatients for Addictive Disorders
Brief Title: Addictology Expert Patients' Fields of Intervention
Acronym: HAPEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP190489
Record Dates: First submitted 2020-01-27; First posted 2020-07-07 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2020-10

CONDITIONS: Substance-Related Disorders
Keywords: expert patients; addictology; withdrawal; addiction
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: patients hospitalized for addiction withdrawal in the addiction service of the university hospital Bichat, Paris, France
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expert patient in addictology (Experimental): before/ after comparison, each patients being its own control
  Interventions: Behavioral: Expert patient in addictology

INTERVENTIONS:
Behavioral: Expert patient in addictology — EP's Intervention, with patients hospitalized for addiction withdrawal. These are weekly individual interviews, in room, proposed by the EPs to inpatients.
  The content of the intervention will be defined trough the results of step one of the study.

SUMMARY:
Although there are many publications concerning the benefit of the interventions of the self-help movements and peer health mediators in psychiatry, no studies have described the intervention specific to patients with expertise in addictology (EP), nor evaluated their effectiveness.

The objective of this study is twofold: identify and define the fields of intervention of EPs adapted to the specific needs of addictology patients. And validate, through a pilot study, the intermediate effectiveness of EP intervention. This EP intervention will be built on the areas of expertise defined in the first step. Intermediate effectiveness will be measured by patients' ability to manage their addiction. The first part of the study will consist of a preliminary qualitative patient-centered study to clarify patients' needs and expectations regarding the content of the EPs' intervention into a one addictology service of the university hospital of Bichat, Paris, France. This will make it possible to translate these needs into fields of expertise to address during the EPs' intervention and will result in the creation of a hetero-questionnaire. The second part of the study will consist of a before-and-after comparative study on inpatients who are their own controls based on the hetero-questionnaire constructed through the qualitative study.

This study will identify the main EP's intervention fields in addictology in which EP are more relevant to patients. Thus, their inpatient interventions can be validated and improved, and better carried by addiction professionals.

DETAILED DESCRIPTION:
1. Targeted population : Major individuals hospitalized in the Department of Addictology and Psychiatry at Bichat Hospital. All participants sign a hospitalization contract upon arrival in which they undertake, among other things, to meet with the EP, within the framework of a system set up in the hospitalization unit since 2015. In order to be able to study the different factors influencing the intervention mechanism, it is decided to take the broadest possible selection criteria in order to remain representative of the heterogeneity of the target population. This is why the investigators have chosen to include all hospitalized patients in the service who agree to meet with an EP, at all socio-economic levels, for withdrawal from any substance regardless of the severity of the addictive disorder, regardless of the previous course of care with or without anxiety and depression symptoms
2. Inclusion criteria : Adults, hospitalized during the period of inclusion of the study in the addictology department at the Bichat-Claude Bernard Hospital in Paris, for withdrawal. Substance use disorder, diagnosed according to the criteria of the DSM-5, i.e. at least 2 diagnostic criteria. Patients who have received information about the research and signed the consent form.
3. Non inclusion criteria : Severe cognitive disorders, i.e. MoCA test < 11, Severe psychiatric disorders assessed using the MINI test (acute psychotic episode, manic or hypomanic episode, severe depression), No understanding of French, Patient under guardianship or curatorship, Patient refusal
4. Study conduct : STEP 1: Preliminary qualitative study

   * among the first eligible patients in the study to specify the content of EP's intervention, adapted to the inpatient's needs
   * Individual face-to-face interview, conducted by the principal investigator (PI) , according to the methodology socio-anthropological interviews
   * The interview will be conducted during the patient's hospitalization, whether the patient has already met with the EP or not.
   * Number of participants expected is not decided, the PI waiting for the saturation of information as it happens as the interviews progressed
   * A semi-structured interview grid will be followed
   * The interviews will be recorded and transcribed in the form of verbatim and then analyzed according to the content analysis technique
   * This analysis will be supervised by a socio- anthropologist from the research team of Robert Debré
   * The needs of patients will be produced by this analysis, and will be translated into fields of skills to be addressed during the EP's intervention
   * End of the study for these first participants

   STEP 2: Before and after comparative study on inpatients being their own witnesses. This is a study feasibility pilot
   * Eligible participants will be patients meeting the criteria for judgment and not having not participated in the first part of the study
   * They will be presented with the study and the collection of the consent at the beginning of hospitalization, before the EP's intervention
   * After agreement of participation, the initial socio-economic participants' characteristics will be collected on the variable collection notebook
   * Completion of the first competency assessment hetero-questionnaire before the EP's intervention (main criterion judgment evaluation). This questionnaire will have been constructed based on patient needs expressed in Part 1
   * EP's Intervention, with patients hospitalized for withdrawal. These are weekly individual interviews, in room, proposed by the EPs to inpatients.
   * The second hetero-questionnaire will be proposed to the same patient during his hospitalization, within 48 hours of the EP's intervention (main criterion judgment evaluation)
   * A follow-up (by telephone or in person) will be carried out at 1 month and then 3 months to estimate the number of patients who have consumed during the hospitalization (frequency, quantity, duration)
   * End of the study for a patient
5. Inclusion : For the qualitative study, the investigators estimate that the data are saturated between 10 and 20 patients. For the quantitative study, the investigators estimate that there are 10 new patients per month. The investigators hope to include at least half of the target population, meaning 50 participants over the 10 months of the study. In total, for the entire study, an estimate of 70 participants.
6. Statistics analysis : The statistical analysis will be performed using SAS v9.3®. The quantitative variables will be presented as median, interquartile and missing data. The qualitative variables will be presented in terms of frequency, percentage and number of missing data. The initial characteristics of the patients will be presented. The indicators qualitative and quantitative acceptability will also be presented. The median of the results of the competency questionnaires between D0 and H48 will be compared between the group before and after by a Wilcoxon test (no hypothesis on the distribution of this variable). A multivariate analysis will be conducted to identify all the factors influencing the variation in questionnaire responses. This will allow the influence of patient profiles on outcomes to be taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the addictology department at the Bichat-Claude Bernard Hospital in Paris, for withdrawal.
* Substance use disorder, diagnosed according to the criteria of the DSM-5, i.e. at least 2 diagnostic criteria.
* Patients who have received information about the research and signed the consent form.

Exclusion Criteria:

* Severe cognitive impairment i.e. MoCA scale < or = 10
* Severe psychiatric conditions assessed using the MINI scale : Acute psychotic episode, Manic or hypomaniacal episode, Severe depression
* non comprehension of french
* patient Under guardianship or curatorship
* patient refusal

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
median of the difference of the score of the competency questionnaires between D0 and H48 will be compared between the group before and the group after | 48 hours
  This EP intervention will be built on the areas of expertise defined in the first step. Intermediate effectiveness will be measured by patients' ability to manage their addiction. This will be measured by a hetero-questionnaire, created by the first part of the study, evaluating the skills acquired by patients before and after this intervention. As this is a new scale created thanks to the forst part of the study, the investigators don't know what will be the minimum, the maximum or/and the relation between the score and the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Chanaëlle OBADIA, MD, Principal Investigator — APHP; Aurélie BOURMAUD, PhD, Study Director — APHP
Locations (1):
- Département psychiatrie et addictologie Bichat Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No